CLINICAL TRIAL: NCT03912376
Title: Feasibility Study of a Hyperspectral Imaging System in Detection of Human Skin Perfusion and Oxygenation
Brief Title: A Study of a Device Used to Take Pictures of Skin Blood Flow
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-098
Record Dates: First submitted 2019-04-08; First posted 2019-04-11 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2024-09

CONDITIONS: Basal Blood Flow
Keywords: Blood Flow; Healthy Participant; Memorial Sloan Kettering Cancer Center; 19-098

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteer: Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history.
  Interventions: Diagnostic Test: Quest Hyperspectral Imaging System

INTERVENTIONS:
Diagnostic Test: Quest Hyperspectral Imaging System — In this camera 3 sensors are combined for optimal spectral imaging. For 2D reference, and to facilitate annotating the data, a high resolution (full HD) color image, recorded with an RGB-sensor, is included with each hyperspectral dataset.

SUMMARY:
The purpose of this study is see fi the hyperspectral camera system (HCS) can measure skin blood flow (perfusion and oxygenation) in healthy people.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, 18 to 45 years of age, inclusive. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history.
* Body mass index (BMI) between 18 to 30 kg/m2, inclusive, and with a minimum weight of 50 kg.
* Able to participate and willing to give written informed consent and to comply with the study restrictions.

Exclusion Criteria:

* History or symptoms of any significant disease including (but not limited to), neurological, psychiatric, endocrine, cardiovascular, respiratory, gastrointestinal, hepatic, or renal disorder.
* Systolic blood pressure (SBP) greater than 140 or less than 90 mm Hg, and diastolic blood pressure (DBP) greater than 90 or less than 50 mm Hg.
* Use of any medications (prescription or over-the-counter [OTC]), vitamin, mineral, herbal, and dietary supplements within 21 days of study drug administration, or less than 5 half-lives (whichever is longer). Exceptions are paracetamol (up to 4 g/day). Other exceptions will only be made if the rationale is discussed and clearly documented between the Investigator and the sponsor.
* Concomitant disease or condition that could interfere with, or for which the treatment of might interfere with, the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this study.
* Smokers as defined by any of the following criteria:
* Reported smoking of cigarettes within 12 months prior to screening; occasionally a cigarette is allowed, but not within 24 hours of the measurement.
* Any confirmed significant allergic reactions (urticarial or anaphylaxis) against any drug, or multiple drug allergies (non-active hay fever is acceptable).
* Unwillingness of inability to comply with the study protocol for any other reason.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Enrollment in this study will be open to all Memorial Sloan Kettering employees to act as healthy volunteers provided they meet eligibility criteria. Every effort will be made to include women and minorities in the research study. Employees who provide consent willfully and voluntarily may participate as a healthy volunteer once.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Bradbury, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Volunteer
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 23.5 [21 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Evaluated to Measure Blood Flow and Oxygenation in the Brachial Artery
Description: Number of participants evaluated to measure blood flow and oxygenation in the brachial artery
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 8
Participants | 8

2. Primary Outcome: Mean Cutaneous Tissue Oxygen Saturation/StO2
Description: Measure changes in blood flow when vessels constrict or dilate by mean measurements Cutaneous Tissue Oxygen Saturation/StO2
Time Frame: Up to 6 months
Measure: Median (Standard Deviation); unit: percentage of StO2
Arm/Group | Healthy Volunteer
Number analyzed (Participants) | 8
percentage of StO2
  Basal Phase | 86.6 (10.0)
  Maximum occlusion | 72.3 (15.9)
  Reperfusion | 85.5 (9.9)

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Healthy Volunteer
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT03912376/Prot_SAP_001.pdf
  • Informed Consent Form (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT03912376/ICF_000.pdf